CLINICAL TRIAL: NCT02852226
Title: Connecting Resources for Urban Sexual Health: CRUSH-PrEP for Women
Brief Title: CRUSH-PrEP for Women Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Gilead Sciences (Industry); Lifelong Medical Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-17574
Record Dates: First submitted 2016-05-10; First posted 2016-08-02 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Sexually Transmitted Diseases; HIV
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Intervention (Experimental): Assess PrEP among women in the study. Assess the characteristics of women who enroll in the PrEP study. Assess the referral sources of women who enroll in the PrEP study
  Interventions: Other: Pre Exposure Prophylaxis; Behavioral: Characteristics of women who enroll; Behavioral: referral sources of women who enroll

INTERVENTIONS:
Other: Pre Exposure Prophylaxis — Uptake will be measured as the proportion of female patients at the LifeLong clinic who are approached that start PrEP after being offered PrEP, the numbers and rate of PrEP discontinuation, the reasons given for PrEP discontinuation (side effects, no longer at risk, fear of stigma, inability to adhere), and drug concentrations. Drug concentrations are monitored using dried blood spots, which have a large dynamic range capable of detecting use of a few pills every month up through daily use. The main measure of PrEP utilization is the proportion of time that PrEP is used effectively among those attempting to use PrEP.
  Other Names: PrEP
Behavioral: Characteristics of women who enroll — The investigators are interested in characterizing the women who decide to take PrEP through this project. Demographic and psychosocial variables will be used to describe the population who enroll. Sexual and behavioral risk profiles of those who decide to initiate PrEP will also be described as part of this study. Demographics of women who uptake PrEP through community partners will also be compared to the demographics of Alameda County women who have incident HIV infection. In addition to demographics and risk behavior, the investigators will also describe the contraceptive use and intentions of women on PrEP towards future pregnancies as these may be important factors driving interest in PrEP among women.
Behavioral: referral sources of women who enroll — Process data will capture the outreach efforts made to recruit participants for this study. At the time of baseline visit, the investigators will capture the source of referral for each woman screened, as well as the primary reason for joining the study. Enrollment progress will be carefully tracked against outreach activities to monitor the relationship between outreach efforts and demand generation. This will help to inform future implementation of PrEP among women.

SUMMARY:
UCSF is conducting an evaluation of a demonstration project. The aims of the CRUSH-PrEP for Women project are to integrate the delivery of a comprehensive PrEP package for HIV-negative at-risk women into primary care settings. The delivery of the PrEP package will leverage the well regarded reputation of the LifeLong primary care clinicians to provide a highly effective combination HIV prevention strategy including; PrEP, post-exposure prophylaxis (nPEP), repeat HIV and STI testing, treatment of sexually transmitted infections. Counselling for for sexual health promotion and services specifically designed for vulnerable women such as staying free of violence and domestic abuse will be offered as an integrated part of this package. UCSF will conduct evaluation activities only. The investigators expect that UCSF will enroll 50 participants in the evaluation assessments across the 15 months of data collection. Evaluation cohort participants will provide quantitative data to evaluate the linkage and engagement in care among clinic attendees as well as the uptake and use of Pre-Exposure Prophylaxis.

DETAILED DESCRIPTION:
The overall goal of the CRUSH PrEP for Women Project is to enhance and extend a response to the local HIV/AIDS epidemic in Alameda County with a set of innovative, evidence-based interventions across the continuum of HIV prevention and care, which target the individuals and communities that are the most vulnerable to HIV infection. The investigators hypothesize that women in Oakland will be interested in accessing PrEP through a community based clinic. Specifically, the CRUSH PrEP for Women Project is a 16month demonstration project designed to evaluate and assess the adherence of PrEP within a community based clinic. The specific aims of the project are as follows:

Aim 1. Assess uptake and adherence to PrEP among women in the study: Uptake will be measured as the proportion of female patients at the LifeLong clinic who are approached that start PrEP after being offered PrEP, the numbers and rate of PrEP discontinuation, the reasons given for PrEP discontinuation (side effects, no longer at risk, fear of stigma, inability to adhere), and drug concentrations. Drug concentrations are monitored using dried blood spots, which have a large dynamic range capable of detecting use of a few pills every month up through daily use. The main measure of PrEP utilization is the proportion of time that PrEP is used effectively among those attempting to use PrEP. Because the effective dose of PrEP is less well characterized for women, only blood concentration levels consistent with daily use will be considered effective use for this analysis. After the supply of study provided medication is ended at 12 months, participants will be followed for an additional 3 months to determine the proportion who continued on PrEP. The investigators will describe patterns of use and the barriers and facilitators to continued use beyond one year. The investigators will look at demographic, and psychosocial and risk factors that may be associated with less than daily adherence to medication, and describe reasons for early discontinuation of PrEP among any women who choose to stop taking medication prior to the end of the first 12 months. Factors associated with discontinuation at the end of the 12-month study provided supply of medication will also be described. Although these analyses will be exploratory, the investigators hypothesize that changes in relationships and pregnancy intentions will be related to changes in PrEP use.

Aim 2. Assess the characteristics of women who enroll in the PrEP study: For Aim 2, the investigators are interested in characterizing the women who decide to take PrEP through this project. Demographic and psychosocial variables will be used to describe the population who enroll. Sexual and behavioral risk profiles of those who decide to initiate PrEP will also be described as part of this study. Demographics of women who uptake PrEP through our community partners will also be compared to the demographics of Alameda County women who have incident HIV infection. In addition to demographics and risk behavior, the investigators will also describe the contraceptive use and intentions of women on PrEP towards future pregnancies as these may be important factors driving interest in PrEP among women.

Aim 3: Assess the referral sources of women who enroll in the PrEP study: Process data will capture the outreach efforts made to recruit participants for this study. At the time of baseline visit, the source of referral for each woman screened will be captured, as well as the primary reason for joining the study. Enrollment progress will be carefully tracked against outreach activities to monitor the relationship between outreach efforts and demand generation. This will help to inform future implementation of PrEP among women.

ELIGIBILITY:
Inclusion Criteria:

* Women who are over 18, able to provide consent in English and intending to reside in the study area for the next 15 months and meeting the eligibility criteria for PrEP per the American College of Obstetricians and Gynecologists 2014 recommendations will be enrolled and complete a baseline evaluation visit.

Eligibility criteria include: women not infected with HIV who are in one or more of the following risk groups:

1. have a male sexual partner who is HIV positive
2. engage in sexual activity within a high HIV-prevalence area or social network, and who have one or more of the following risk factors:

   Inconsistent or no condom use,

   Diagnosis of sexually transmitted infections,

   Exchange of sex for commodities,

   Use of intravenous drugs or alcohol dependence or both,
3. have sexual partners of unknown HIV status with any of the factors previously listed.

Exclusion Criteria:

* Absolute Exclusion Criteria:

  * Under the age of 18
  * Inability to provide informed consent in English
  * Intention to leave the study area within the following 15 months
  * Insufficient renal function (estimated creatinine clearance less than 60 mL/min)
  * HIV infected
  * Breastfeeding

Potential Exclusion Criteria:

* High risk known or suspected exposure to HIV within 72 hours prior to presentation;
* Osteoporosis;
* History of pathological bone fractures not related to trauma;
* Ongoing therapy with a drug with significant nephrotoxic potential (other than over the counter non-steroidal anti-inflammatory drugs taken as directed);
* Concomitant participation in a clinical trial using investigational agents, including placebo-controlled clinical trials using such agents;
* Any other conditions that are deemed contraindications for PrEP by the NP/MD; or
* Any other condition that would preclude provision of informed consent; make participation in the project unsafe; complicate interpretation of outcome data; or otherwise interfere with achieving the project objectives, based on the opinion of the investigators and/or treating clinician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The proportion of women eligible for PrEP who choose to access PrEP. | 1 year
Monitor adherence to PrEP through pharmacy pick up information. Self reported adherence and blood levels. | 48 weeks
  Pharmacy records will be accessed to monitor pick-up records. Self administered quantitative interviews will collect self reported adherence to PrEP. Dried blood spot tests are conducted to establish the amount of PrEP taken.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Myers, PhD, Principal Investigator — UCSF Center for AIDS Prevention; Mi-Suk Kang Dufour, PhD, Principal Investigator — UCSF Center for AIDS Prevention; Kimberly A Koester, MA, Principal Investigator — UCSF Center for AIDS Prevention; Rebecca Packard, BA, Study Director — UCSF Center for AIDS Prevention
Locations (1):
- Lifelong Medical Care, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Access is restricted to those who successfully submit a protocol to the UCSF IRB.

REFERENCES:
- [Background] Eisingerich AB, Wheelock A, Gomez GB, Garnett GP, Dybul MR, Piot PK. Attitudes and acceptance of oral and parenteral HIV preexposure prophylaxis among potential user groups: a multinational study. PLoS One. 2012;7(1):e28238. doi: 10.1371/journal.pone.0028238. Epub 2012 Jan 11. PMID 22247757
- [Background] Gupta N, Schmidt H, Buisker T, Dufour MS, Goldenson J, Myers J, Tulsky J. After the Fact: A Brief Educational Program on HIV Postexposure Prophylaxis for Female Detainees in a Local Jail. J Correct Health Care. 2015 Apr;21(2):140-51. doi: 10.1177/1078345815572335. PMID 25788609
- [Background] Koester KA, Maiorana A, Vernon K, Myers J, Rose CD, Morin S. Implementation of HIV prevention interventions with people living with HIV/AIDS in clinical settings: challenges and lessons learned. AIDS Behav. 2007 Sep;11(5 Suppl):S17-29. doi: 10.1007/s10461-007-9233-8. Epub 2007 Apr 11. PMID 17436072
- [Result] Auerbach JD, Kinsky S, Brown G, Charles V. Knowledge, attitudes, and likelihood of pre-exposure prophylaxis (PrEP) use among US women at risk of acquiring HIV. AIDS Patient Care STDS. 2015 Feb;29(2):102-10. doi: 10.1089/apc.2014.0142. Epub 2014 Dec 16. PMID 25513954